CLINICAL TRIAL: NCT05857228
Title: Epigenetic Modulation Drives Chronic Type 2 Chronic Rhinosinusitis With Nasal Polyposis: Identifying Markers, Pathogens and Mechanisms
Brief Title: Viral and Epigenetic Influences in CRSwNP
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 08.149
Record Dates: First submitted 2023-05-02; First posted 2023-05-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: CRSwNP; Epigenetic; Virus; Infection; Microbiome
MeSH Terms: conditions — Disease; Virus Diseases; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, nasal biopsies and/or nasal brushings
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary epithelial cells: Population: The investigators will use frozen dissociated cells from our biobank in earliest possible format (P0 or P1) to preserve original viruses and epigenetic marks. Polyp samples from T2 CRSwNP will be selected according to clinical phenotype together with blood test and histology.
- Patients in remission of CRSwNP: Population: Perfect sinus cavity outcome after ESS under continued intranasal corticosteroids (INCS) or dupilumab.
- Effect of sinus surgery on the sinus virome: Population: Patients undergoing ESS for CRSwNP, including at least 30% of subjects with aspirin sensitivity.
  Interventions: Procedure: Endoscopic sinus surgery (ESS)
- Healthy volonteers: Population: Participants with no sino-nasal symptoms and normal sense of smell as assessed by UPSIT-40 testing.

INTERVENTIONS:
Procedure: Endoscopic sinus surgery (ESS) — Endoscopic sinus surgery for removal of nasal polyps and sinus tissue.
  Groups: Effect of sinus surgery on the sinus virome

SUMMARY:
Background/rationale

While multiple disorders feature a Type 2 (T2) inflammation, triggers for T2 remains unknown. In Chronic Rhinosinusitis with Nasal Polyposis CRSwNP), a classic Type 2 disorder, dysfunction of the epithelial barrier is suggested by loss of epithelial cell differentiation, impaired response to wounding, and impairment of innate defense mechanisms. After unsuccessful attempts to describe T2 disorders solely by host genetic or environmental factors, the role of epigenetics in the modification of innate immune response and epithelial integrity appears an important unexplored mechanism for a novel appreciation of T2 disease.

In addition, the investigators explore the possibility that these changes may be induced by viral pathogens. This concept has been supported by the recent observation that SARS-CoV-2 viral reduction measures resulted in a reduction of the frequency of respiratory viruses and a concomitant reduction in chronic airway disease, suggesting a role for viruses in T2 disease.

Hypothesis

The investigators believe T2 chronic rhinosinusitis (CRSwNP) involves epigenetic mechanisms where external factors, possibly viruses, contribute to disease via epigenetic manipulation and/or chronic viral infection.

Objectives

The investigators aim to identify epigenetic signatures associated with T2 CRS and explore the contribution of viruses. Method A robust methylation profiling with extensive coverage will be used for epigenome-wide association studies in T2 CRS patients assessing healthy subjects, CRS patients in remission, and diseased patients undergoing surgery. Moreover, advanced transcriptomic and metagenomic methods will identify gene expression profiles and viruses. This proposal also includes a cross-sectional study of patients undergoing surgery to assess transcriptomic patterns and epigenetics at the single-cell level.

Expected outcome

The investigators expect to identify epigenetic biomarkers and implicate several pathogenic viruses to open new targets for novel therapies.

DETAILED DESCRIPTION:
RESEARCH BACKGROUND & RATIONALE

Chronic rhinosinusitis (CRS) can manifest as T2 and/or non-T2 inflammation patterns, independently of the presence or absence of nasal polyps (NP). Certain aspects of CRS, such as NP formation, have been associated with epigenetic processes. Numerous studies support a role for epigenetics in the development and chronicity of other T2 diseases e.g. asthma and allergic rhinitis (North, Ann Allergy Asthma Immunol, 2011).

An insight into T2 disease pathogenesis may have been afforded by the "real-world" experiences during the COVID19 pandemic. Viral containment measures deployed in 2020 predictably reduced the frequency of most common respiratory viruses, reducing invasive respiratory infections along with exacerbations of asthma and COPD, which are typically triggered by viral respiratory infections (Linden, Eur Respir Rev, 2019; Mikhail, Ann Allergy Asthma Immunol, 2019). Unexpectedly, chronic inflammation of the upper airways was also reduced. Chronic otitis media with effusion and adenoiditis plummeted, and over half of the children on the waiting list for surgery the investigators removed because of spontaneous improvement. This was accompanied by anecdotal observations of a reduction in consultations for chronic rhinosinusitis with nasal polyposis (CRSwNP).

The investigators thus propose that T2 disease represents a unique facet of the inflammatory disease spectrum whereby dysfunction develops following interaction with a viral pathogen maintaining persistent effects via epigenetic mechanisms or chronic infection.

Detailed Research Plan Current understanding of T2 disease pathophysiology leaves early steps of pathogenesis largely unexplained. The investigators believe T2 disease is a result of epigenetic imprinting which reduces T1 response to injury or pathogens via impairment of Interferon (IFN) signaling components, leading to unopposed T2 signaling.

Furthermore, the investigators suspect that this dysfunction is produced by viral infection, which may persist in the host in latent form, or which may continue to exert its effects via epigenetic modifications of the host genome. In consequence, the investigators propose to comprehensively characterize the epigenetic modulations present in T2 inflammation, with a focus on demonstrating the link with viral infections. To reach our goal, the investigators will characterize T2 disease by combining DNA methylation status, chromatin accessibility and gene expression profiling to determine genes and epigenetic changes potentially important in the pathogenesis of T2 disease. The investigators will leverage the massive change in societal viral exposure imposed by pandemic measures as a unique experimental condition by comparing contemporary results with a biobank of pre- pandemic material. In addition to shedding new light on the pathogenesis, defining the epigenetic and virome portrait of T2 disease will improve new diagnostic and therapeutic targets, and potentially, identify implicated viruses.

Research strategy The investigators will identify epigenetic patterns and viruses associated with T2 CRSwNP patients . Taking advantage of an existing and extensive biobank of cells from tissue and biopsy samples, the investigators will compare epigenetics and viruses present pre-lockdown and per- pandemic in CRS and healthy patients. The population (detailed in the next section) includes healthy subjects, CRS patients under treatment in remission, and diseased patients undergoing endoscopic sinus surgery (ESS). The investigators aim to assess an equal number of both biological sexes to analyse potential differences. Sample size is based on previous transcriptomics experience. This observational study will not require any additional treatment to patients.

Experimental design

I) TYPE 2 AND METHYLATION:

Primary epithelial cells from CRSwNP biopsy samples (N=24) and control primary nasal epithelial cells from patients undergoing endoscopic pituitary surgery (N=16) Population: The investigators will use frozen dissociated cells from our biobank in earliest possible format (P0 or P1) to preserve original viruses and epigenetic marks. Polyp samples from T2 CRSwNP will be selected according to clinical phenotype together with blood test and histology.

II) PATIENTS IN REMISSION Methods: Experiments A, B and C will all use the following method for analysing brushing samples from the nasal cavity. (N=36) A) Establishing the virome and methylation profile in healthy upper airway cells. (N=12) B) What do healthy sinuses look like under medical treatment (N=12) C) Does reducing T2 inflammation with dupilumab work by increasing IFN activity or by reducing methylation in IFN pathway?

III) HOW DOES SURGERY EXERT AN EFFECT ON TYPE 2? Primary cross-sectional analysis and then compared to evolution at 4 months post-surgery Population: Patients undergoing ESS for CRSwNP, including at least 30% of subjects with aspirin sensitivity.

Phase I: At time of ESS (n= 24, plus 6 for validation of brushing) Methods: Patients will undergo a biopsy of the anterior ethmoid sinus. These will be undergo assessment using transcriptomic tools, including Single cell multiomes .

Phase II: 4 months post-ESS (n=the same 24 paired subjects. The same cohort of patients will be assessed at the four-month timepoint. Evolution of disease will be assessed according to CSO HNS standards into "Optimal" "Sub-optimal" or "Unacceptable" results. A brushing will be used for sampling and subjected to the same analyses as above.

ELIGIBILITY:
Inclusion Criteria:

* T2 CRSwNP patients with favorable evolution
* T2 CRSwNP patients undergoing ESS
* Healthy volonteers with no nasal symptoms and documented normal sense of smell

Exclusion Criteria:

* Cystic fibrosis
* Primary immunodefisciencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * T2 CRSwNP patients with favorable evolution
  * T2 CRSwNP patients undergoing ESS
  * Healthy volonteers with no nasal symptoms and documented normal sense of smell
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Identification of epigenetic biomarkers and pathogenic viruses | 12 months
  The investigators expect to identify viruses and epigenetic markers associated with CRS.
  Viruses will be identified using bulk sequencing of collected tissue. Viruses will be considered "present" only if they are seen on at least 5 reads in sequencing. These identified viruses will be considered as associated with disease or healthy states assessed only when they are seen in at least 25% of tissue samples for the given condition. Association with disease will be defined as a higher proportion of candidate virus in diseased as opposed to healthy conditions.
  Epigenetic markers will be identified by comparing methylation profiles across the whole genome between active CRSwNP disease with disease in remission. Machine learning techniques will be used to identify putative sequences of epigenetic biomarkers associated with active disease or presence of an identified viral pathogen.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Y. Desrosiers, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] North ML, Ellis AK. The role of epigenetics in the developmental origins of allergic disease. Ann Allergy Asthma Immunol. 2011 May;106(5):355-61; quiz 362. doi: 10.1016/j.anai.2011.02.008. Epub 2011 Mar 16. PMID 21530865
- [Background] Linden D, Guo-Parke H, Coyle PV, Fairley D, McAuley DF, Taggart CC, Kidney J. Respiratory viral infection: a potential "missing link" in the pathogenesis of COPD. Eur Respir Rev. 2019 Mar 14;28(151):180063. doi: 10.1183/16000617.0063-2018. Print 2019 Mar 31. PMID 30872396
- [Background] Mikhail I, Grayson MH. Asthma and viral infections: An intricate relationship. Ann Allergy Asthma Immunol. 2019 Oct;123(4):352-358. doi: 10.1016/j.anai.2019.06.020. Epub 2019 Jul 2. PMID 31276807